CLINICAL TRIAL: NCT03639519
Title: 'A Prospective Randomized Trial to Assess the Impact of Ascorbic Acid on Outcomes and Complications Post Cardiac Surgeries''
Brief Title: A Trial to Assess the Impact of Ascorbic Acid on Cardiac Surgeries Outcomes and Complications''
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: El-Galaa Military Medical Complex (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMMC-RC18-2
Record Dates: First submitted 2018-08-13; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Cardiothoracic Surgery
MeSH Terms: interventions — Ascorbic Acid; Mastication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ascorbic acid (Experimental): Patients will take 2 g orally ascorbic acid effervescent tablets the night before cardiac surgery, then 1 g twice daily for 5 days after surgery in addition to their traditional medical care.
  Interventions: Drug: Ascorbic Acid 500Mg Chew Tab
- Placebo group (Placebo Comparator): will not be given ascorbic acid , instead a placebo will be used, and will be given the rest of traditional medical care provided to the first arm. Inflammatory markers (CRP, ESR and differential TLC), serum urea and creatinine, ALT, AST, CK-mb, CK-Total, aPTT, INR, Hemoglobin, platelet count, will be assessed on day 0, 1,2,4,6 postoperative in both arms.
  Interventions: Other: Carbonated orange beverage

INTERVENTIONS:
Drug: Ascorbic Acid 500Mg Chew Tab — Ascorbic acid will be administered at the night before surgery and will be continued for five days
  Arms: Ascorbic acid
Other: Carbonated orange beverage — The carbonated orange beverage will be administered at the night before surgery and will be continued for five days
  Arms: Placebo group

SUMMARY:
this study is evaluating the safety and efficacy of ascorbic acid as a drug that can decrease inflammatory complications post surgical in addition to its impact on decreasing risk of arrhythmia and total opioid administration post operative

DETAILED DESCRIPTION:
The study will include two arm of patients who are scheduled for elective cardiac surgery, either coronary artery bypass grafting (CABG) or Valvular replacement First arm: Patients will take 2 g orally ascorbic acid effervescent tablets the night before cardiac surgery, then 1 g twice daily for 5 days after surgery in addition to their traditional medical care. Second arm: will not be given ascorbic acid , instead a placebo 9orange carbonated beverage) will be used, and will be given the rest of traditional medical care provided to the first arm. Inflammatory markers C- reactive protein (CRP), erythrocyte sedimentation rate (ESR) and differential total leukocytic count (TLC), serum urea and creatinine, ALT, AST, CK-mb, CK-Total, aPTT, INR, Hemoglobin, platelet count, will be assessed on day 0, 1,2,4,6 postoperative in both arms.

ELIGIBILITY:
Inclusion Criteria:

* Elective Cardiac surgery
* American Society of Anesthesiologists physical status class I-III

Exclusion Criteria:

* Allergy to ascorbic acid
* Asthma
* COPD
* Allergy to opioids
* Previous history of chemical dependence
* Prior cardiac surgery
* Known hyperoxaluria
* History of renal calculi
* History of allergic or hypersensitivity reaction to ascorbic acid products
* Currently taking 1 g or more of ascorbic acid supplementation daily

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-04-15 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Risk of arrhythmia post operative | 7 days post operative
  assessing risk of AF post surgical using ECG
pain management | 2 days post operative
  Evaluating cumulative dose of opioid administered within ICU stay in the two groups
wound healing | 30 days post operative
  assessment of wound inflammation and infection risk using ASEPSIS score (a scoring system to assess wound healing and evaluate the presence of infection, a score between 10 to 20 means disturbed healing, >20 points means infected wound, >30 means moderate to sever infection)

CONTACTS AND LOCATIONS:
Locations (1):
- Galaa Military Medical Complex, Cairo, Sheraton, Egypt